CLINICAL TRIAL: NCT06887361
Title: The Efficacy of a New Sexual Violence Prevention Program with College Students: a Randomized Controlled Trial
Brief Title: Evaluating the Efficacy of a New Sexual Violence Prevention Program with College Students
Acronym: MOON Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: University of Coimbra (Other); Aveiro University (Other); Foundation for Science and Technology, Portugal (Other); Center for Psychology at the University of Porto, Portugal (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MOONProgram; 2022.12638.BD (Other Grant/Funding Number: Foundation for Science and Technology)
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Sexual Violence
Keywords: Clinical trial; Sexual Violence; Prevention; College Students; Bystander Approach

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Participants allocated to this arm will receive intervention (i.e., will participate in the MOON sessions).
  Interventions: Behavioral: MOON Program
- Control Group (No Intervention): Participants allocated to this arm will be part of a control group, not receiving intervention and participating exclusively in the assessment time points.

INTERVENTIONS:
Behavioral: MOON Program — The MOON Program aims to contribute to the primary prevention of sexual violence among young university students. The program aims to achieve this goal by promoting bystander attitudes and behaviors through psychoeducation and skills training that enable participants to be active agents in this process. During the sessions, beliefs that legitimize violence will be deconstructed and skills such as communication about consent and empathy will be promoted. The MOON program consists of five online sessions, which are intended to be completed autonomously on a weekly basis. Throughout the sessions, participants will learn on the following topics: SV and consent, gender stereotypes, SV myths and bystander attitudes and behaviors.
  Arms: Experimental Group

SUMMARY:
This research project will develop, deliver, and assess the efficacy of a new sexual violence (SV) prevention program for college students. The MOON program (Moving ON against sexual violence) aims to prevent sexual violence amongst university students, who are known to be an at-risk population for this form of violence.

The MOON program follows a bystander approach, aiming to teach and capacitate young adults to be active agents of prevention within their communities. To do so, the program combines education on several SV-related topics with skills-training activities.

Throughout five online sessions, the participants will be educated on topics such as sexual violence and consent, gender stereotypes, SV myths and bystander attitudes and behaviors. The main goal is to promote discussion forums, increase the participants knowledge on these topics and deconstruct pre-conceived beliefs/ideas that promote societal tolerance and acceptance of SV The program follows a bystander approach to support young adults in the development of bystander attitudes and behaviors that will help them act in situations of risk of SV. To achieve this goal, the program sessions will also have a major focus on building bystander prevention skills through online practical exercises (e.g., training scenarios).

Finally, the program also focuses on promoting empathy towards others, specifically in the context of sexual violence prevention. This focus aims to deconstruct victim blaming narratives and to build victim-support skills, to enhance the students' sense of responsibility and their proclivity to act and help others in need. Being empathic towards others is perceived as a crucial component in the bystander decision-making to intervene.

This clinical trial will apply the MOON program with university students nationwide in the Portuguese context and compare the participants who will take part in the program (experimental group) with other students who will not (control group). Thus, the RCT will be conducted with the following goals:

1. To assess the treatment's efficacy, by evaluating the program's ability to significantly reduce gender stereotypes, sexism, and rape myths; and to significantly increase active bystander attitudes and behaviors and empathy towards other people.
2. To examine the extent to which any changes are maintained three, six and nine months after the program's completion.
3. To assess mechanisms of change, i.e., to test whether changes in cognitive outcomes, namely in rape myth endorsement, are associated with changes over time in behavioral outcomes, as bystander attitudes/behaviors.
4. To investigate the role of age and gender as moderators of change over time in SV perpetration, gender stereotypes, sexism, rape myths, bystander attitudes and behaviors and empathy.

DETAILED DESCRIPTION:
Project Relevance:

Literature places evidence of consistently high rates of SV perpetration among university populations, highlighting the need to design prevention programs that target specifically this type of violence in this population. The delivery of the MOON program fits within the framework of human rights established internationally in the Istanbul Convention and aligns with the World Health Organization's recommendation of major focus on primary prevention for SV.

Design and Participants:

The present project consists of a randomized controlled trial (RCT). The study will be conducted following the guidelines by the CONSORT-SPI Group.

This project follows a longitudinal design. Participants will answer a set of self-report measures in five different time-points: one week before the beginning of the program (baseline), one week after the program's completion (post-test), and three, six and nine months after the post-test (follow-up assessments).

Power analysis showed that a sample of 179 participants will be necessary to detect medium effects with a significance level of .05 and a power of .95. The sample will include a minimum of 200 male and female participants. Inclusion criteria require participants to be 18 years old or older, to be fluent in the Portuguese language and to be attending college.

Inclusion criteria:

Participants must be 18 years old or older. All participants must be enrolled in a higher education institution in Portugal. Finally, participants will have to be fluent in written and spoken Portuguese.

Intervention:

MOON (MOving ON against sex violence) is a SV prevention program for college students. The MOON is an online program of five sessions which are meant to be completed autonomously on a weekly basis. To promote the development of active bystander attitudes and behaviors on the participants, they will be educated and complete different exercises on the following topics along the sessions: SV and consent, gender stereotypes, SV myths, empathy and bystander attitudes and behaviors.

The contents of each session are as follow:

1. Sexual Violence (Framing SV as a public health matter; informing about SV and its various forms and contexts it can occur in; and teaching about the importance of recognizing consented vs. non-consented sexual interactions.)
2. Pro-Social Attitudes (Defying myths and beliefs that promote tolerance to SV; understanding the barriers to the bystander intervention vs. learning strategies to overcome those barriers; and promoting the participants' pro-social attitudes.)
3. Empathy (Promoting empathy towards others; fostering the participants' sense responsibility to act; and introducing the role of the active bystander in the prevention of SV.)
4. Pro-Social Behaviors (Promoting pro-social bystander behaviors of the participants; and sharing and training practical examples of bystander intervention in SV incidents)
5. Bystander Skills (Training practical intervention skills and preparing the participants to be active agents of SV prevention).

Measures To assess the intended outcomes, several self-report measures will be combined into a survey: Bystander Attitudes and Behaviors Scales; three items to measure Empathy Social; Rape Myth Scale; Social Role Questionnaire; Inventory of Ambivalent Sexism and Desirability Scale.

Procedures According to the statistical power analysis, approximately 200 university students will be recruited. This study will be advertised through university mailing lists and on social media platforms. The program objectives and contents will be presented to the participants, and the research will follow upon informed consent. Students who voluntarily agree to participate in the study will start by completing the online self-report survey (evaluating gender stereotypes, sexism, SV myths endorsement, bystander attitudes and behaviors and empathy) on the week prior to the intervention (baseline). Due to the self-report nature of the measurements, a social desirability measure will also be included to control for potential bias of the participants responses. Afterwards, individual randomization of participants to each group (control and intervention) will be ensured using a randomization software (https://www.randomizer.org/). Each condition will include approximately 100 participants. This distribution accounts for possible and expected dropouts and ineligible participants. Students assigned to the intervention group will then complete the programs' sessions online during five weeks. Remaining participants will be assigned to the wait list control group. Students of both experimental conditions will also answer the survey at the post-test assessment (the week after the programs' completion) and at the three, six- and nine-months follow-ups. The moderator factors (age and gender) will be assessed exclusively at baseline. The programs' integrity will be ensured through: (a) specific intervention manual, (b) ongoing supervision of the process, and (c) direct assessment of the participants' adherence throughout the five weeks.

Data analysis:

All analysis will be carried out according to an intention-to-treat analysis. To assess treatment outcomes in the completers, a per-protocol analysis will also be carried out. Treatment and moderator effects will be analyzed Unconditional and Conditional Latent Growth Models. To examine mechanisms of change, two-wave latent change scores models will be performed. All analyses will be done through Mplus v.8.7.

ELIGIBILITY:
Inclusion Criteria:

18 years old or older Enrolled in a Portuguese university Fluent in Portuguese (written and spoken)

-

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Bystander Attitudes | Assessed at five different timepoints: (1) baseline - one week prior to the beginning of the program, (2) post-test - one week after the completion of the program and (3-5) follow-ups of three, six and nine months counting from the post-test assessment.
  Bystander attitudes - Bystander Attitudes Scale - Revised (BAS-R) assesses bystander attitudes in SV scenarios (e.g., "Confront a friend if I hear rumors that they had forced someone to have sex"). For each scenario, participants are asked to indicate to what extent the described is acceptable according to a 5-point Likert scale that ranges from (1) = "Not acceptable" to (5) = "Extremely Acceptable". This instrument originally consisted of a 4-factor model categorizing items/scenarios by (1) High-risk Situations, (2) Post-assault Support for the Victim; (3) Post-assault Reporting of the Perpetrator; and (4) Proactive Opportunities. The Portuguese version of the measurement consists of 14 items organized into three similar subdimensions: (1) High-risk Situations, (2) Victims Support/Protection Behaviors, and (3) Proactive Opportunities.
Bystander Behaviors | Assessed at five different timepoints: (1) baseline - one week prior to the beginning of the program, (2) post-test - one week after the completion of the program and (3-5) follow-ups of three, six and nine months counting from the post-test assessment.
  Bystander behaviors - Bystander Behaviors Scale - Revised (BBS-R) assesses bystander behaviors within SV scenarios through 16 self-report items (e.g. "Say something to a friend who is taking a drunk person back to their room at a party"). For each scenario participants are asked if they ever been in the described situation and the response varies across "Yes", "No" and "I haven't been in that situation". The original measurement instrument is organized by a 2-factor model contemplating (1) Intervention Opportunities and (2) Proactive Opportunities.

SECONDARY OUTCOMES:
Empathy | Assessed at five different timepoints: (1) baseline - one week prior to the beginning of the program, (2) post-test - one week after the completion of the program and (3-5) follow-ups of three, six and nine months counting from the post-test assessment.
  Empathy - Empathy is to be measured with three items (see Milfont & Sibley, 2016). The items correspond to different affirmations (i.e., "I sympathize with others' feelings"; "I am not interested in other people's problems," reversed score; "I feel others' emotions"). Participants are asked to indicate their agreement with each statement accordingly to a seven-point Likert-type scale ranging from 1 (Strongly Disagree) to 7 (Strongly Agree).
Myths about sexual violence | Assessed at five different timepoints: (1) baseline - one week prior to the beginning of the program, (2) post-test - one week after the completion of the program and (3-5) follow-ups of three, six and nine months counting from the post-test assessment.
  Myths about sexual violence will be assed with the sexual violence myths Scale. The scale assesses the subject's degree of tolerance/acceptance of the use of SV. The items are organized into five different factors that allow a better understanding of the specific beliefs underlying the tolerance to SV. The measurement includes items such as "Some people deserve to be raped" and "Some people get sexual pleasure when they are raped". Participants are asked to rate their agreement to each statement accordingly to a Likert scale ranging from 1 ("Completely Disagree") to 5 ("Completely Agree").
Attitudes about gender roles | Assessed at five different timepoints: (1) baseline - one week prior to the beginning of the program, (2) post-test - one week after the completion of the program and (3-5) follow-ups of three, six and nine months counting from the post-test assessment.
  Gender role attitudes - Social Role Questionnaire (SRQ) assesses attitudes toward social roles. The scale includes items such as "People can be both aggressive and nurturing regardless of sex"; "Men are more sexual than women"; and "Mothers should work only if necessary." Respondents are asked to indicate how much they agree with each item by choosing a percentage range that varies between 0% and100%, with increments of 10%.
Sexism | Assessed at five different timepoints: (1) baseline - one week prior to the beginning of the program, (2) post-test - one week after the completion of the program and (3-5) follow-ups of three, six and nine months counting from the post-test assessment.
  Sexism - Inventory of Ambivalent Sexism (IAS) allows the identification of beliefs related to sexist practices, including the sub scale of hostile sexism (i.e., more visible sexual discrimination - e.g. "Women are too easily offended") and the sub scale benevolent sexism (i.e., more subtle pejorative attitudes - e.g. "Women, compared to men, tend to have a superior moral sensibility"). The responses vary within in a Likert scale from 1 ("Completely Disagree") to 5 ("Completely Agree").
Social Desirability | Assessed at five different timepoints: (1) baseline - one week prior to the beginning of the program, (2) post-test - one week after the completion of the program and (3-5) follow-ups of three, six and nine months counting from the post-test assessment.
  Social Desirability Scale - EDS-20 assesses behaviors and attitudes considered socially desirable, involving the denial of negative characteristics and the attribution of positive qualities through 20 dichotomous response items ("Yes" / "No").

CONTACTS AND LOCATIONS:
Overall Officials: Joana Carvalho, PhD, Study Director — William James Research Center, Department of Education and Psychology, University of Aveiro
Locations (1):
- University of Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almiro PA, Marques PRF, Duarte MC, Alberto IM, Simoes MR. Validation study of the Roberts Apperception Test for Children (RATC) in an adolescents' forensic sample. Acta Psychol (Amst). 2023 May;235:103900. doi: 10.1016/j.actpsy.2023.103900. Epub 2023 Mar 31. PMID 37004420
- [Background] Jouriles EN, Krauss A, Vu NL, Banyard VL, McDonald R. Bystander programs addressing sexual violence on college campuses: A systematic review and meta-analysis of program outcomes and delivery methods. J Am Coll Health. 2018 Aug-Sep;66(6):457-466. doi: 10.1080/07448481.2018.1431906. Epub 2018 Mar 12. PMID 29405865
- [Background] Martins, S., Machado, C., Abrunhosa, R., & Manita, C. (2012). Escala de Crenças sobre Violência Sexual (ECVS). Análise Psicológica, 30(1 / 2), 177-191. https://doi.org/10.14417/ap.546
- [Background] McMahon S, Allen CT, Postmus JL, McMahon SM, Peterson NA, Lowe Hoffman M. Measuring bystander attitudes and behavior to prevent sexual violence. J Am Coll Health. 2014;62(1):58-66. doi: 10.1080/07448481.2013.849258. PMID 24313697
- [Background] Grant S, Mayo-Wilson E, Montgomery P, Macdonald G, Michie S, Hopewell S, Moher D; , on behalf of the CONSORT-SPI Group. CONSORT-SPI 2018 Explanation and Elaboration: guidance for reporting social and psychological intervention trials. Trials. 2018 Jul 31;19(1):406. doi: 10.1186/s13063-018-2735-z. PMID 30060763
- [Background] Mikton C. Preventing intimate partner and sexual violence against women: taking action and generating evidence. Inj Prev. 2010 Oct;16(5):359-60. doi: 10.1136/ip.2010.029629. No abstract available. PMID 20921563
- [Background] Kettrey HH, Marx RA. The Effects of Bystander Programs on the Prevention of Sexual Assault across the College Years: A Systematic Review and Meta-analysis. J Youth Adolesc. 2019 Feb;48(2):212-227. doi: 10.1007/s10964-018-0927-1. Epub 2018 Sep 27. PMID 30264210
- [Background] Katz J, Moore J. Bystander education training for campus sexual assault prevention: an initial meta-analysis. Violence Vict. 2013;28(6):1054-67. doi: 10.1891/0886-6708.vv-d-12-00113. PMID 24547680
- [Background] Krug EG, Mercy JA, Dahlberg LL, Zwi AB. The world report on violence and health. Lancet. 2002 Oct 5;360(9339):1083-8. doi: 10.1016/S0140-6736(02)11133-0. PMID 12384003
- [Background] Carvalho J, Rosa PJ, Pereira B. Dynamic Risk Factors Characterizing Aggressive Sexual Initiation by Female College Students. J Interpers Violence. 2021 Mar;36(5-6):2455-2477. doi: 10.1177/0886260518760010. Epub 2018 Mar 5. PMID 29502500
- [Background] Carvalho J, Sa A. Male College Students Using Sexually Aggressive Strategies: Findings on the Interpersonal Relationship Profile. J Interpers Violence. 2020 Feb;35(3-4):646-661. doi: 10.1177/0886260516689779. Epub 2017 Jan 30. PMID 29294637
- [Background] McDaniel MC, Rodriguez DN. Undergraduate Men's Self-Reports of Sexual Assault and Perceptions of College Campus Acquaintance Rape. J Interpers Violence. 2021 Feb;36(3-4):1772-1790. doi: 10.1177/0886260517743552. Epub 2017 Nov 29. PMID 29295008
- [Background] Krahe B, Berger A. Men and women as perpetrators and victims of sexual aggression in heterosexual and same-sex encounters: a study of first-year college students in Germany. Aggress Behav. 2013 Sep-Oct;39(5):391-404. doi: 10.1002/ab.21482. Epub 2013 Apr 29. PMID 23629691